CLINICAL TRIAL: NCT00222885
Title: Three-Tracer PET Quantitation of Insulin Action in Muscle
Brief Title: Multi-Tracer PET Quantitation of Insulin Action in Muscle (Phase 1, Phase 2, Phase 3, Phase 4)
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Other Study IDs: 011178; R01DK060555 (NIH)
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2007-12-19 (Estimated); Status verified 2007-12

CONDITIONS: Diabetes; Obesity
Keywords: PET imaging; Skeletal muscle; In vivo insulin-stimulated tissue perfusion; Glucose transport; Glucose phosphorylation
MeSH Terms: conditions — Diabetes Mellitus; Obesity

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The purpose of this research is to develop a new method to study insulin action using positron emission tomography (PET). Insulin is the hormone made by your body to control the blood sugar level. We want to develop a way to image (look at) the following three things: 1) how insulin affects blood flow in skeletal muscle 2) how insulin affects glucose (sugar) transport (movement) into muscle, and 3) how insulin affects glucose metabolism (breakdown) in skeletal muscle of healthy individuals. The long term goal will be to later apply this method to the study of metabolic diseases, especially type 2 diabetes mellitus and obesity.

PET imaging is a relatively non-invasive way to obtain a "metabolic picture" of body organs, and has been used successfully to study brain, heart and more recently skeletal muscle. In this research study, we will use PET with as many as four radioactive tracers (markers) to study skeletal muscle glucose transport in healthy volunteers.

DETAILED DESCRIPTION:
The goal of this proposal is to develop a novel triple-tracer positron emission tomography (PET) method to image in vivo insulin-stimulated tissue perfusion, glucose transport and glucose phosphorylation in skeletal muscle in healthy individuals. The long term goal will be to later apply this model to the study of metabolic diseases, notably type 2 diabetes mellitus (Type 2 DM) and obesity (Ob). While it is often suggested that glucose transport is the rate-controlling step for insulin action, we will test the hypothesis that the control insulin exerts on the uptake of glucose into skeletal muscle is distributed across flow and tissue perfusion, trans-membrane transport and intra-cellular phosphorylation of glucose.

Specific Aim 1. The first specific aim is to develop the triple-tracer PET method for quantitative determinations of tissue perfusion, glucose transport and glucose phosphorylation in skeletal muscle. To measure blood flow and tissue perfusion, we will use 15O-H2O (half-life ~ 2 min; also referred to as 15O-water). To measure glucose transport, we will use 11C-3-O-methyl glucose (half-life ~ 20 min; also referred to as 3-0-MG), an analog that is transported but not phosphorylated or otherwise metabolized. 18F-2-deoxy-2-fluoro-glucose (half-life ~ 109 min; also referred to as FDG), will be used to examine glucose transport and glucose phosphorylation. Because of the differences in half-life of the three positrons (15O, 11C, and 18F), it is feasible to use each of these tracers, in sequence, in the same individual.

Specific Aim 2. The second specific aim is to rigorously test mathematical models to extract quantitative physiological information from dynamic PET imaging. We will test a novel model that specifically addresses the kinetics of substrate delivery within the interstitial space of skeletal muscle (i.e. a 5 rate constant, 4 compartment model with respect to FDG. Model testing will entail use of non-compartmental models e.g. spectral analysis).

ELIGIBILITY:
Inclusion Criteria:

* We will recruit normal weight (BMI 19 to 25 kg/m2), glucose tolerant, healthy volunteers, who are between the ages of 20 and 45 years old. Volunteers for this study must have a fasting glucose < 100 mg/dl; HbA1c < 6.0; Hct > 34; ALT < 60; AST < 60; Alk phos < 150; TSH < 8; Trig < 300; Chol < 250; systolic BP < 150; diastolic BP < 95; negative family history (first-degree relatives) for type 2 DM; be in good health and not be taking any chronic medications. Previous difficulty with xylocaine will be an exclusion. To be eligible for these studies, volunteers must be free of clinical evidence of cardiac, renal, hepatic, and vascular disease, or other major medical problems that would endanger the volunteers or compromise the scientific validity of the studies. Subjects with a history of myocardial infarction, proteinuria (defined as 1+ protein), liver disease, alcohol or drug abuse, malignancy or neuromuscular disease will be excluded.

Exclusion Criteria:

* Subjects will be excluded if taking chronic medications known to adversely affect glucose homeostasis including thiazide diuretics, oral glucocorticoids, nicotinic acid, and beta-blockers. Subjects who have gained or lost more than 3 kg during the past 6 months will be excluded. Because of the PET scanning, all premenopausal women must have a negative pregnancy test within 24 hours prior to these procedures and this will be confirmed prior to each PET scanning session. These subjects will also be advised to use reliable contraceptive techniques during the study period. To avoid radiation exposure of the infant, women who are currently breastfeeding will not be permitted to participate in this research study. Subjects participating in Phase 2 and Phase 4 (that includes an MRI Scan) will be excluded if they have a contraindication to MRI such as surgical or vascular implants, pregnancy, pacemaker, or claustrophobia. In subjects with a questionable history of metallic fragments, an X-ray of the suspected area of the body will be performed to rule such out.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50
Dates: Start 2002-12; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Triple tracer PET method development for in vivo imaging of skeletal muscle metabolism

SECONDARY OUTCOMES:
Testing of mathematical modeling of PET data

CONTACTS AND LOCATIONS:
Overall Officials: David E Kelley, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Result] Bertoldo A, Price J, Mathis C, Mason S, Holt D, Kelley C, Cobelli C, Kelley DE. Quantitative assessment of glucose transport in human skeletal muscle: dynamic positron emission tomography imaging of [O-methyl-11C]3-O-methyl-D-glucose. J Clin Endocrinol Metab. 2005 Mar;90(3):1752-9. doi: 10.1210/jc.2004-1092. Epub 2004 Dec 21. PMID 15613423